CLINICAL TRIAL: NCT02930122
Title: A Prospective, Single-Center, Randomized, Triple-Blinded, Placebo-Controlled Study of IL-1RA Treatment in Patients With Acute ACL Tear and Painful Effusions
Brief Title: IL-1RA Treatment in Patients With Acute ACL Tear and Painful Effusions
Acronym: EASI ACL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Cale Jacobs, PhD (Other)
Responsible Party: Sponsor-Investigator, Cale Jacobs, PhD, Assistant Professor Research, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 45595
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anakinra (Experimental): Intervention: anakinra (150mg) Participants will receive an intraarticular injection of anakinra (150mg) at 0-28 days post injury
  Interventions: Drug: anakinra (150mg)
- Placebo Control (Placebo Comparator): Intervention: Saline (0.9%) Participants will receive a saline placebo injection within 28 days of injury
  Interventions: Other: Saline intraarticularly

INTERVENTIONS:
Drug: anakinra (150mg) — intraarticular administration
  Other Names: Kineret
  Arms: Anakinra
Other: Saline intraarticularly — intraarticular administration
  Other Names: Saline (0.9%)
  Arms: Placebo Control

SUMMARY:
Injury to the knee during sports participation often involves partial or full detachment of the anterior cruciate ligament (abbreviated as ACL). ACL tears cause pain, swelling and inflammation. While the swelling and inflammation usually goes away in time, individuals with ACL injuries may experience pain and notice knee instability (knee slipping, etc.). Often surgery can repair or replace the ACL within the joint, allowing individuals the ability to walk or run again pain free or participate in sports. Unfortunately, osteoarthritis of the knee, which also causes pain and swelling, can occur in that same knee 10-20 years later for reasons which are not well understood.

In this research study, the investigator hopes to reduce the initial pre-operative pain. The reduction of pain will allow for earlier movement of the knee joint and preparation for surgery. The investigator is interested to see if the use of Kineret does decrease the risk of developing arthritis in individuals with ACL injuries by treating them within 28 days after their injury.

DETAILED DESCRIPTION:
Kineret® was chosen because it is safe, well tolerated, and has been used to treat Rheumatoid Arthritis (RA) and post-surgical persistent knee effusions as well as knee stiffness. Although Kineret® is approved by the US Food and Drug Administration (FDA) for the treatment of RA and Neonatal-Onset Multisystem Inflammatory Disease, it is not currently approved by the FDA for use in treating ACL injury. Therefore, the use of Kineret® in this study is investigational.

The research procedures will be conducted at the University of Kentucky (UK) Medical Center. Participants will need to come to the UK Healthcare at Turfland located at 2195 Harrodsburg Road in Lexington, KY. Participants will be asked to come to this location seven times during the study. Each of those visits will take about 30 minutes. All exams and questionnaires will be administered during the otherwise necessary routine visits for any participant who has suffered an ACL tear. No additional visit is necessary. The total amount of time commitment for participation in this study is about 6 1/2 hours, over the next 2 years.

All participants with sports related ACL injuries enrolled in this study will be seen and may elect to undergo surgery, if necessary. Note: Surgery is not part of this protocol. Should participants be enrolled into the study and choose not to undergo ACL reconstruction (surgery), they will receive treatment according to this protocol.

Randomization: Once it has been determined that a participant qualifies for entry into the study, they will be randomized, like the flipping of coin into one of two treatment groups. Groups will receive knee injections with either Kineret® or a saline placebo. The saline placebo will contain no active medication. Both the participant and study doctor will not know what treatment group the participant is assigned to. However, in case of an emergency, the investigator will be able to find out what treatment group the participant has been assigned to.

* Group 1 will receive an injection of Anakinra (Kineret®, IL-1ra; 150mg) 1-28 days after ACL injury.
* Group 2 is the placebo group. Participants enrolled into this group will receive an injection of saline placebo at Visit 1.

X-rays: All participants would have undergone a routine clinical x-ray analysis at prior to Visit 1.

MRI: All participants will undergo initial MRI examination to confirm ACL injury at Visit 1 and subsequent MRIs will be performed at Visits 5 and 6.

Participants will undergo knee aspirations. During a knee aspiration, the investigator will remove fluid from the space around the knee using a needle and syringe. This is usually performed under a local anesthetic to either relieve swelling or to obtain fluid for analysis to diagnose a joint disorder and/or problem. Knee aspirations after ACL tear with a painful effusion are a common orthopaedic practice and standard of care in at the UK Medical Center. Thus they are not considered additional interventions with regard to this study unless the participant has no fluid in the knee.

At Visit 1: Participants may have a large effusion that requires aspiration. This would be done as part of the participants normal routine care.

At Visit 2: Should the participant elect to undergo ACL reconstruction surgery, they will undergo a study required knee aspiration. This will be performed for the purpose of the research.

At Visit 3: Should the participant elect to undergo ACL reconstruction surgery, and there is substantial post-operative fluid in the knee, the investigator may choose to aspirate the knee again. This would be done as part of the participants normal routine care.

After the aspiration procedure: Once home, it is important for the participant to keep the joint aspiration site clean and dry. The aspiration site may be tender or sore for a few days after the joint aspiration procedure. The investigator will instruct the participant on what pain reliever they may take.

Below is breakdown of what will happen at each study visit:

Visit 1 Screening (1-28 days following injury)

* Obtain informed consent and assent if necessary of potential subjects
* Review medical history to determine eligibility based on inclusion/exclusion criteria.
* MRI scheduled
* Review medications history to determine eligibility based on inclusion/exclusion criteria.
* Perform medical examinations and collect vital signs as needed to determine eligibility based on inclusion/exclusion criteria. All subjects must have a clinical exam that is consistent with an ACL tear.
* Height and weight will be recorded
* Collection of urine and blood for laboratory testing. Women of child bearing potential will be given a urine pregnancy test. Test must be negative in order to enroll into the study. Parents/Legal Guardians of minor females: Your child will have a pregnancy test to see if they are eligible to be in the study. The results will not be disclosed to anyone other than your child, except in the case of a risk to health or welfare.
* Subjects will have the following assessments: range of motion, knee instability (Lachman's test) and standardized weight bearing x-rays. At this time the subjects will also be asked to fill in a standard questionnaire covering the KOOS, IKDC, VR-12, and a Likert pain scale.

Following the review of above assessment results and a review of inclusion/exclusion criteria, subjects will be randomized into 1 of 2 treatment groups. Following randomization, subjects will undergo a knee aspiration and will receive their first dose study medication.

Visit 2 (day of surgery or 4-6 weeks post injury)

* Medical history
* Medication history
* ROM will be performed
* Knee aspiration (in the operating room under anesthesia. This will be omitted if you do not have surgery)
* KOOS, IKDC, VR-12, and a Likert pain scale administered prior to surgery
* Biomarkers (urine and serum) pre-operatively
* Review AEs and SAEs

Visit 3 (4-14 days after Visit 2)

* Knee aspiration (if clinical indicated)
* Biomarkers (urine and serum)
* Review for AE's and SAE's
* ROM will be performed

Visit 4 (6 months after Visit 2)

* Patient reported outcomes (PROs) administered
* KOOS, IKDC, VR-12, and a Likert pain scale administered
* ROM will be performed
* Review of AEs and SAEs

Visit 5 (12 months after Visit 2)

* MRI
* Patient reported outcomes (PROs) administered
* KOOS, IKDC, VR-12, and a Likert pain scale administered
* Biomarkers (serum and urine only)
* Review of AEs and SAEs
* ROM will be performed

Visit 6 (24 months after Visit 2)

* MRI
* Patient reported outcomes (PROs) administered
* KOOS, IKDC, VR-12, and a Likert pain scale administered
* Biomarkers (urine and serum)
* Review of AEs and SAEs
* ROM will be performed

The blood and fluid samples collected from the participants will NOT UNDERGO GENETIC TESTING. Samples will be analyzed and stored at a UK research laboratory. The will be tested for special markers of cartilage breakdown and will remain property of the University of Kentucky indefinitely or until they are completely used. The results from the analyzed samples are important only for research For this reason, these results will not be released to either the participant or their family.

Either the participant or their insurance company, Medicare or Medicaid will be responsible for the costs of all care and treatment they receive during this study that they would normally receive for their condition.

The University of Kentucky may not be allowed to bill an insurance company, Medicare or Medicaid for the medical procedures done strictly for research. These costs include the following:

* X-ray of the knee done at Visit 1
* Knee aspiration done at Visit 1 and Visit 3 (if necessary)

The University of Kentucky may not be allowed to bill your insurance company, Medicare or Medicaid for the medical procedures done strictly for research. The following will be provided at no cost to you: the injection of Kineret®, the second knee aspiration and potentially the third knee aspiration, questionnaires and three MRIs.

Participants will receive $150.00 for taking part in this study. They will receive $50.00 for each MRI completed. Payment will be in the form of a check which will be mailed approximately four to six weeks following the study visit. If the participant is a child the compensation will be mailed to the child.

Should a participant decide to withdraw from the study early they will be compensated for their time and travel.

ELIGIBILITY:
Inclusion Criteria:

* Acute ACL Tear and Painful Effusions
* Signed and dated combined informed consent/HIPAA form and if a minor, a signed assent.
* Willingness to comply with all study procedures and availability for the duration of the study
* For females of reproductive potential: use of highly effective contraception.
* Currently participating in a sporting activity
* Documentation of closed growth plates as noted on the screening x-ray

Exclusion Criteria:

* underlying inflammatory disease (i.e. Rheumatoid Arthritis, Psoriatic Arthritis etc)
* have been diagnosed with hepatitis B or tuberculosis
* currently have an infections, including infection of the skin, or have signs and symptoms of an infection, including fever.
* any abnormalities in their white blood cell counts
* have a disease that weakens your immune system such as diabetes, cancer, HIV or AIDs
* other major medical condition requiring treatment with immunosuppressant or modulating drugs.
* A history of chronic use of non-steroidal anti-inflammatory drugs
* Currently taking immunosuppressant medication, including oral and parenteral corticosteroids (topical and stable dose inhaled corticosteriods are acceptable)
* Females who are pregnant or breastfeeding
* Received a "live" vaccine (smallpox, MMR (measles, mumps and rubella), flu, polio, typhoid, chicken pox, yellow fever, herpes zoster) 4 weeks prior to screening.
* A history of bleeding disorders or are taking any blood thinning medications, aspirin or other medications affecting blood clotting.
* Previous exposure or allergic reaction to anakinra
* Allergy to latex or tape
* Allergy to Kineret or have had a reaction to any local or general anesthesia
* prior knee surgery (contralateral)
* have received any investigational drug with 4 weeks of study Visit 1

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Austin Stone, MD, Study Chair — University of Kentucky
Locations (1):
- UK Healthcare at Turfland, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An insufficient number of participants were consented to generate meaningful data for this study as the study was terminated due to lack of funding.
Period: Overall Study
Arm/Group | Anakinra | Placebo Control
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — The trial was terminated prior to participating completing the study due to lack of funding. | 3 | 3

BASELINE CHARACTERISTICS:
Population: 6 participants had been enrolled at the time the study was closed (3 participants in each group)
Groups:
- Arm 1: Intervention: anakinra (150mg) Participants will receive an intraarticular injection of anakinra (150mg) at 0-28 days post injury
  anakinra (150mg): intraarticular administration
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Placebo Control | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 16 [16 to 17] | 18 [14 to 21] | 17 [14 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptom Score [Median (Full Range); unit: units on a scale] — KOOS symptoms scores range from 0 to 100, with higher scores indicating less severe symptoms.
  units on a scale | 14 [10 to 16] | 15 [11 to 15] | 14.5 [10 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Change of Knee Injury and Osteoarthritis Outcome Score (KOOS) Symptom Score Between Groups
Description: KOOS symptoms scores range from 0 to 100, with higher scores indicating less severe symptoms.
Time Frame: 1 year
Population: The trial was terminated due to lack of funding so an insufficient number of participants were consented to generate meaningful data.
Arm/Group | Arm 1 | Placebo Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in CTX-II Levels From Injury to Time of Surgery
Description: CTX-II levels measured by ELISA
Time Frame: time of surgery
Population: as for outcome 1
Arm/Group | Anakinra | Placebo Control
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: MRI T1rho Changes
Description: MRI: T1rho values in Medial and lateral femoral condyle as well as medial and lateral tibial plateau
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Anakinra | Placebo Control
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) Score Between Groups
Description: KOOS QOL
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Anakinra | Placebo Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm 1 | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT02930122/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02930122/ICF_001.pdf